CLINICAL TRIAL: NCT03054545
Title: Evaluation of Clinical Efficacy and Immunologic Response After Iguratimod Therapy in Refractory Lupus Nephritis
Brief Title: Iguratimod as Treatment for Refractory Lupus Nephritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: [2017]27
Record Dates: First submitted 2017-02-11; First posted 2017-02-15 (Actual); Last update posted 2017-02-27 (Actual); Status verified 2017-02

CONDITIONS: Lupus Nephritis
MeSH Terms: conditions — Lupus Nephritis | interventions — iguratimod; T 614

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Iguratimod treating group (Experimental): Iguratimod 25mg twice a day, oral administrated.
  Interventions: Drug: Iguratimod

INTERVENTIONS:
Drug: Iguratimod — Iguratimod 25mg twice a day, oral administrated.
  Other Names: T-614

SUMMARY:
This study is to evaluate the efficacy and safety of a novel chemical synthetic agent iguratimod as treatment of refractory lupus nephritis. All subjects should have at least one failed immunosuppressive treatment and suffer active nephritis at the screening stage. The study period is 52 week. All the subject will receive therapy of iguratimod combined with steroids.

ELIGIBILITY:
Inclusion Criteria:

* Active lupus nephritis:

Fulfill ACR classification criteria (2009) for SLE Proteinuria ≥1g/24h at screening stage experience at least one failed therapy within one year before screening, including but not limit to cyclophosphamide, methotrexate, azathioprine, mycophenolate mofetil, cyclosporin, tacrolimus and leflunomide. The regime can be monotherapy or combination. Any regime should be at least applied for six months.

* Body weight ≥40kg
* SLE-2K score ≥8
* Agreement of contraception
* Informed consent obtained

Exclusion Criteria:

* Active severe SLE-driven renal disease or unstable renal disease at screening
* Active severe or unstable neuropsychiatric SLE
* Clinically significant active infection including ongoing and chronic infections
* History of human immunodeficiency virus (HIV)
* Confirmed Positive tests for hepatitis B or positive test for hepatitis C
* Active tuberculosis
* Live or attenuated vaccine within 4 weeks prior to screening
* Subjects with significant hematologic abnormalities
* Abnormal liver function test at screening (ALT, AST or total bilirubin over 2 fold of upper normal level
* History of peptic ulcer or GI bleeding; treatment with warfarin or other anticoagulants within last 14 days

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-05-08 (Estimated); Primary Completion 2018-05-08 (Estimated); Study Completion 2019-04-30 (Estimated)

PRIMARY OUTCOMES:
Renal remission rate | Week 52

SECONDARY OUTCOMES:
Renal remission rate | Week 24
Renal flare rate | Week 52
Number of participants with treatment-related adverse events | Week 52
  Adverse events are assessed by CTCAE v4.0
Systemic Lupus Erythematosus Disease Activity Index inSafety of Estrogens in Lupus Erythematosus National Assessment (SELENA-SLEDAI) | Week 52
British Isles Lupus Activity Group (BILAG) score | Week 52
PGA | Week 52
  Patient general assessment
Quality of life | Week 52
  Measured by HAQ

CONTACTS AND LOCATIONS:
Locations (1):
- RenJi Hospital, Shanghai, Shanghai Municipality, China